CLINICAL TRIAL: NCT03358706
Title: A Phase 1, Open-label, Drug Interaction Study to Evaluate the Effect of Ustekinumab on Cytochrome P450 Enzyme Activities Following Induction and Maintenance Dosing in Participants With Active Crohn's Disease or Ulcerative Colitis.
Brief Title: A Study to Evaluate the Effect of Ustekinumab on Cytochrome P450 Enzyme Activities Following Induction and Maintenance Dosing in Participants With Active Crohn's Disease or Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped as all post-marketing commitments had been fulfilled or released
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108352; CNTO1275CRD1003 (Other: Janssen Research & Development, LLC); 2017-000831-16 (EudraCT Number)
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Crohn Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Midazolam; Warfarin; Vitamin K; Omeprazole; Dextromethorphan; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crohn's Disease or Ulcerative Colitis Participants: Ustekinumab + Probe Cocktail (Experimental): Participants will receive a single Intravenous (IV) infusion dose of ustekinumab (dosage to be decided based on body weight) on Day 8 and a ustekinumab 90 milligram (mg) maintenance dose via subcutaneous (SC) route on Day 64. A second optional maintenance dose may be administered on Day 120 based on participants clinical response assessed by investigator. The probe cocktail (2 milligram [mg] of midazolam, 10 mg of warfarin plus 10 mg of vitamin K, 20 mg of omeprazole, 30 mg dextromethorphan, and 100 mg of caffeine) will be administered orally on Days 1, 22, and 113.
  Interventions: Drug: Ustekinumab IV Infusion; Drug: Ustekinumab SC Injection; Drug: Midazolam 2 mg; Drug: Warfarin 10 mg; Drug: Vitamin K 10 mg; Drug: Omeprazole 20 mg; Drug: Dextromethorphan 30 mg; Drug: Caffeine 100 mg
- Healthy Participants: Probe Cocktail (Experimental): Participants will receive the probe cocktail (2 mg of midazolam, 10 mg of warfarin plus 10 mg of vitamin K, 20 mg of omeprazole, 30 mg dextromethorphan, and 100 mg of caffeine) orally on Day 1.
  Interventions: Drug: Midazolam 2 mg; Drug: Warfarin 10 mg; Drug: Vitamin K 10 mg; Drug: Omeprazole 20 mg; Drug: Dextromethorphan 30 mg; Drug: Caffeine 100 mg

INTERVENTIONS:
Drug: Ustekinumab IV Infusion — Participants will receive a single IV infusion dose of ustekinumab (dosage to be decided based on body weight) on Day 8.
  Arms: Crohn's Disease or Ulcerative Colitis Participants: Ustekinumab + Probe Cocktail
Drug: Ustekinumab SC Injection — Participants will receive a Ustekinumab 90 mg SC maintenance dose on Day 64. A second optional maintenance dose may be administered on Day 120 based on participants clinical response assessed by investigator.
  Arms: Crohn's Disease or Ulcerative Colitis Participants: Ustekinumab + Probe Cocktail
Drug: Midazolam 2 mg — Participants will receive 2 milligram per milliliter (mg/ml) syrup of midazolam as a component of the Cytochrome P 450 probe cocktail orally.
Drug: Warfarin 10 mg — Participants will receive 10 mg tablet of warfarin as a component of the Cytochrome P 450 probe cocktail orally.
Drug: Vitamin K 10 mg — Participants will receive 10 mg tablet of vitamin K as a component of the Cytochrome P 450 probe cocktail orally.
Drug: Omeprazole 20 mg — Participants will receive 20 mg capsule of omeprazole as a component of the Cytochrome P 450 probe cocktail orally.
Drug: Dextromethorphan 30 mg — Participants will receive 30 mg capsule of dextromethorphan as a component of the Cytochrome P 450 probe cocktail orally.
Drug: Caffeine 100 mg — Participants will receive 100 mg tablet of caffeine as a component of the Cytochrome P 450 probe cocktail orally.

SUMMARY:
The purpose of this study is to evaluate the potential effects of an intravenous (IV) induction and subcutaneous (SC) maintenance administration of ustekinumab on the pharmacokinetic (PK) of a cocktail of representative probe substrates of cytochrome P450 (CYP) enzymes (CYP3A4, CYP2C9, CYP2C19, CYP2D6, and CYP1A2) in participants with Active Crohn's disease (CD) or Ulcerative Colitis (UC).

ELIGIBILITY:
Inclusion Criteria For Crohn's Disease (CD) Participants

* Participant must have a body weight in the range of 45 to 110 kilogram (kg) inclusive and have a body mass index (BMI) of 18 to 35 kilogram per meter square (kg/m^2) inclusive
* Have had moderate to severe CD or fistulizing CD of at least 3 months duration, with colitis, ileitis, or ileocolitis, confirmed at any time in the past by histology, and/or endoscopy

For Healthy Volunteers

* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Healthy on the basis of clinical laboratory tests performed at screening and Day-1
* If a woman of childbearing potential, she must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at screening; and a negative urine pregnancy test at Day -1

Exclusion Criteria For CD Participants

* Has complications of CD such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation that might be anticipated to require surgery in the next 3 months, could preclude the use of the Crohn's Disease Activity Index (CDAI) to assess response to therapy, would possibly confound the ability to assess the effect of treatment with ustekinumab, or would alter the absorption of the probe cocktail
* Currently has or is suspected to have an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks prior to baseline, or 8 weeks prior to baseline for intra-abdominal abscesses, provided that there is no anticipated need for any further surgery. Participants with active fistulas may be included if there is no anticipation of a need for surgery and there are currently no abscesses identified

For Healthy Volunteers Participants

* Has an abnormal C-reactive protein (CRP) greater than (>) 2* upper limit of normal (ULN)
* Has had major surgery (example, requiring general anesthesia) within 8 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is in screening or is expected to participate in the study (5 weeks)
* Is pregnant, nursing, or planning a pregnancy (both men and women) during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
For Crohn's disease (CD) or Ulcerative Colitis (UC) Participants: Geometric Mean Ratio (Day 22/ Day 1) of the Maximum Plasma Concentration (Cmax) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Day 1 and 22: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  Cmax is defined as maximum observed plasma concentrations. The geometric mean ratio of Cmax will be defined as the Cmax of probe substrates on Day 22/Cmax of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 113/ Day 1) of the Cmax of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Day 1 and 113: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  Cmax is defined as maximum observed plasma concentrations. The geometric mean ratio of Cmax will be defined as the Cmax of probe substrates on Day 113/Cmax of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 22/ Day 1) of the Area Under the Plasma Concentration-time Curve From 0 to Infinity (AUC [0-inf]) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Day 1 and 22: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  (AUC [0-inf]) is defined as area under the plasma concentration versus time curve from time 0 to infinity with extrapolation of the terminal phase. The geometric mean ratio of Cmax will be defined as the (AUC [0-inf]) of probe substrates on Day 22/(AUC [0-inf]) of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 113/ Day 1) of AUC (0-inf) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Day 1 and 113: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  (AUC [0-inf]) is defined as area under the plasma concentration versus time curve from time 0 to infinity with extrapolation of the terminal phase. The geometric mean ratio of (AUC [0-inf]) will be defined as the (AUC [0-inf]) of probe substrates on Day 113/(AUC [0-inf]) of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 22/ Day 1) of Area Under the Plasma Concentration-time Curve From 0 to Last Time (AUC [0-last]) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Day 1 and 22: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  (AUC [0-last]) is defined as the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration. The geometric mean ratio of (AUC [0-last]) will be defined as the (AUC [0-last]) of probe substrates on Day 22/(AUC [0-last]) of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 113/ Day 1) of AUC (0-last) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Day 1 and 113: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  (AUC [0-last]) is defined as the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration. The geometric mean ratio of (AUC [0-last]) will be defined as the (AUC [0-last]) of probe substrates on Day 113/(AUC [0-last]) of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 22/ Day 1) of the Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC [0-24]) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, and Caffeine) | Day 1 and 22: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  (AUC [0-24]) is defined as area under the plasma concentration-time curve from time 0 to 24 hours. The geometric mean ratio of (AUC [0-24]) will be defined as the (AUC [0-24]) of probe substrates on Day 22/(AUC [0-24]) of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 113/ Day 1) of the Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC [0-24]) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, and Caffeine) | Day 1 and 113: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post dose
  (AUC [0-24]) is defined as area under the plasma concentration-time curve from time 0 to 24 hours. The geometric mean ratio of (AUC [0-24]) will be defined as the (AUC [0-24]) of probe substrates on Day 113/(AUC [0-24]) of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 22/ Day 1) of the Area Under the Plasma Concentration-time Curve From 0 to 96 Hours (AUC [0-96]) of Cytochrome P450 Probe Substrate (S-warfarin) | Day 1 and 22: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post dose
  (AUC [0-96]) is defined as area under the plasma concentration-time curve from time 0 to 96 hours. The geometric mean ratio of (AUC [0-96]) will be defined as the (AUC [0-96]) of probe substrates on Day 22/(AUC [0-96]) of probe substrates on Day 1.
For CD or UC Participants: Geometric Mean Ratio (Day 113/ Day 1) of the Area Under the Plasma Concentration-time Curve From 0 to 96 Hours (AUC [0-96]) of Cytochrome P450 Probe Substrate (S-warfarin) | Day 1 and 113: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours post dose
  (AUC [0-96]) is defined as area under the plasma concentration-time curve from time 0 to 96 hours. The geometric mean ratio of (AUC [0-96]) will be defined as the (AUC [0-96]) of probe substrates on Day 113/(AUC [0-96]) of probe substrates on Day 1.

SECONDARY OUTCOMES:
CD and UC Participants: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 (only for dextromethorphan and S-warfarin), 72 (only for S-warfarin) and 96 hours (only for S-warfarin) on Days 1, 22, and 113 postdose administration of cytochrome P450 probe substrates
  Tmax is defined as time to reach the maximum observed plasma concentration of Cytochrome P450 Probe Substrates.
CD and UC Participants: Terminal Half-Life (T1/2) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 (only for dextromethorphan and S-warfarin), 72 (only for S-warfarin) and 96 hours (only for S-warfarin) on Days 1, 22, and 113 postdose administration of cytochrome P450 probe substrates
  T1/2 is defined as the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
CD and UC Participants: Apparent Total Systemic Clearance (CL/F) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 (only for dextromethorphan and S-warfarin), 72 (only for S-warfarin) and 96 hours (only for S-warfarin) on Days 1, 22, and 113 postdose administration of cytochrome P450 probe substrates
  CL/F after extravascular administration is defined as the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
CD and UC Participants: Apparent Volume of Distribution (Vz/F) of Cytochrome P450 Probe Substrates (Midazolam, Omeprazole, Dextromethorphan, S-warfarin and Caffeine) | Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 (only for dextromethorphan and S-warfarin), 72 (only for S-warfarin) and 96 hours (only for S-warfarin) on Days 1, 22, and 113 postdose administration of cytochrome P450 probe substrates
  Vz/F based on terminal phase after extravascular administration is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after subcutaneous dose (Vz/F) is influenced by the fraction absorbed.
CD and UC Participants: Twelve Hour Urine Dextromethorphan to Dextrorphan Ratio | Pre-dose and for 12 hours after probe cocktail administration on Day 1, 22 and 113
  Urine samples will be analyzed to determine 12 hour urine dextromethorphan to dextrorphan ratio.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to Day 176
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were events between administration of study drug and up to Day 176 that were absent before treatment or that worsened relative to pre-treatment state.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (16):
- United States (3):
  - WCCT Global, LLC, Cypress, California
  - Ocean Blue Medical Research Center Inc., Miami Springs, Florida
  - Duke University, Durham, North Carolina
- Belgium (4):
  - Ghent University Hospital, Ghent
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
  - Az Sint-Maarten, Mechelen
  - Clinical Pharmacology Unit, Merksem
- Germany (6):
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - CTC North GmbH & Co. KG, Am Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Clinical Research Center Hannover, Hanover
  - University Hospital Heidelberg, Heidelberg
- United Kingdom (3):
  - Wythenshawe Hospital, Greater Manchester
  - Royal Liverpool University Hospital, Liverpool
  - Guy's Hospital, London